CLINICAL TRIAL: NCT00450983
Title: Transplantation of Haploidentical CD34+ Purified Peripheral Blood Stem Cells With NK-Cell Add-Back Following Conditioning With Total Body Irradiation, Thiotepa, Fludarabine and OKT3
Brief Title: Donor Peripheral Stem Cell Transplant and Donor Natural Killer Cell Transplant After Total-Body Irradiation, Thiotepa, Fludarabine, and Muromonab-CD3 in Treating Patients With Leukemia or Other Blood Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Ann Woolfrey, Principal Investigator, Fred Hutchinson Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: 1965.00; R01AI053193 (NIH); P30CA015704 (NIH); FHCRC-1965.00; CDR0000533834 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: graft versus host disease; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Muromonab-CD3; fludarabine phosphate; Methotrexate; Thiotepa; Gene Expression Profiling; Flow Cytometry; Immunologic Techniques; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: muromonab-CD3
Biological: natural killer cell therapy
Drug: fludarabine phosphate
Drug: methotrexate
Drug: thiotepa
Genetic: gene expression analysis
Other: flow cytometry
Other: immunologic technique
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell and donor natural killer cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When certain stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Removing the T cells from the donor cells before transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving a donor peripheral stem cell transplant and a donor natural killer cell transplant after total-body irradiation, thiotepa, fludarabine, and muromonab-CD3 works in treating patients with leukemia or other blood diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of haploidentical donor CD34+ purified peripheral blood stem cells and donor natural killer (NK) cells on the risk of developing grades III-IV acute graft-vs-host disease in patients with leukemia or other hematologic diseases.

Secondary

* Determine the risk for mortality from infection before day 180 in patients treated with this regimen.
* Determine the risk for graft rejection in patients treated with this regimen.
* Determine the risk for life-threatening infections in patients treated with this regimen.
* Determine the concentration of subsets of NK, NK-T, T cells, and dendritic cells in the CD34+ NK/NK-T-enriched graft.
* Determine cytomegalovirus-specific T-cells in product and donor graft.
* Determine the genotype and phenotype of donor killer cell immunoglobulin-like receptor expression according to time after hematopoietic stem cell transplantation (HSCT).
* Determine the reconstitution of NK function according to time after HSCT.
* Determine the expression of NKG2 ligands of leukemic blasts.

OUTLINE: Patients are stratified according to age (≤ 7 years vs > 7 years).

* Conditioning regimen: Patients 7 years of age or younger undergo total-body irradiation (TBI) twice daily on days -11 to -9. Patients over 7 years of age undergo TBI once on day -9. All patients receive thiotepa IV over 2 hours on days -8 and -7, fludarabine phosphate IV on days -6 to -3 and muromonab-CD3 on days -6 to 6. Patients with acute lymphoblastic leukemia or leukemia in the spinal fluid also receive methotrexate intrathecally prior to and after donor peripheral blood stem cell (PBSC) transplantation .
* Donor PBSC transplantation: Patients undergo donor PBSC transplantation comprising CD34+ purified PBSCs and natural killer (NK) cells on day 0.

Blood samples are collected in weeks 1-4, 6, 8, and 12. Analysis of samples includes quantitation of NK, NK-T, and T-cell subsets (CD3, CD4, and CD8) by flow cytometry; donor killer cell immunoglobulin-like receptor genotype and phenotype; interferon-gamma levels; and NK cytotoxicity. Samples are also analyzed by leukemic blast assay to determine if ligands that activate NK cells are expressed.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following life-threatening hematological malignancies:

  * Acute lymphoblastic leukemia meeting 1 of the following criteria:

    * Advanced beyond first remission
    * In first remission with high-risk prognostic features, including any of the following:

      * Philadelphia chromosome-positive disease
      * Chromosome 11q23 abnormality
      * Hypodiploid
      * Failed to achieve first remission within 1 month after induction
  * Acute myeloid leukemia (AML) meeting 1 of the following criteria:

    * Advanced beyond first remission
    * First remission with high-risk prognostic features, including any of the following:

      * Chromosome 11q23 abnormality
      * Chromosome del 7q
      * Secondary AML
      * Failed to achieve first remission within 1 month after induction
  * Myelodysplastic syndromes with International Prognostic Score > 1
  * Chronic myelogenous leukemia in accelerated or blastic phase
* No active CNS disease
* No suitable HLA-matched related or unrelated donor available
* Haploidentical family member available as donor of partially HLA-matched peripheral blood stem cells

  * Least degree of mismatch to HLA-A, B, C, DRB1, and DQB1
  * No mismatch for a single HLA-A, B, C, DRB1, or DQB1 antigen
  * Donor killer cell immunoglobulin-like receptor ligand group expression preferably different than patient

PATIENT CHARACTERISTICS:

* LVEF ≥ 45%
* DLCO ≥ 60% of predicted
* AST and ALT ≤ 2 times upper limit of normal (ULN) (unless due to malignancy)
* Bilirubin ≤ 2 times ULN (unless due to malignancy)
* No life expectancy < 6 months due to coexisting disease other than the malignancy
* No active infection (e.g., polymerase chain reaction [PCR] evidence for cytomegalovirus, human herpes virus 6, or invasive fungal infection)
* No prior infections without evidence of resolution by PCR or imaging studies within the past 2 months
* No hypersensitivity to murine antibodies
* No known HIV positivity
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior marrow transplantation with total body irradiation > 400 cGy
* No concurrent therapies for seizure disorder
* No growth factors for 21 days after transplantation

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2006-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, MD, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Following total-body irradiation, thiotepa, fludarabine, and muromonab-CD3, participants are given a donor peripheral stem cell transplant and a donor natural killer cell transplant.
Period: Overall Study
Arm/Group | Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 1.7 [1.7 to 1.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Risk of Developing Grades III-IV Acute Graft-vs-host Disease (GVHD)
Description: Count of participants with acute GVHD grades III-IV.
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Risk for Mortality From Infection Before Day 180
Description: Count of participant deaths from infection up to day 180.
Time Frame: Up to day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Risk for Graft Failure
Description: Count of participant that had graft failure.
Time Frame: Engraftment documented day +20
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Risk for Life-threatening Infections
Description: Count of participants with life-threatening infections
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Concentration of NK, NK-T, T-cells, and Dendritic Cell Subsets in the CD34+ NK/NK-T-enriched Graft
Time Frame: Up to 5 years
Population: Analysis for this endpoint not feasible due to funding constraint.
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Cytomegalovirus-specific T Cells in Product and Donor Graft
Time Frame: Up to 5 years
Population: Analysis for this endpoint not feasible due to funding constraint.
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Genotype and Phenotype of Donor Killer Cell Immunoglobulin-like Receptor Expression According to Time After Hematopoietic Stem Cell Transplantation (HSCT)
Time Frame: Up to 5 years
Population: Analysis for this endpoint not feasible due to funding constraint.
Arm/Group | Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Reconstitution of NK Function According to Time After HSCT
Time Frame: Up to 5 years
Population: Analysis for this endpoint not feasible due to funding constraint.
Arm/Group | Treatment
Number analyzed (Participants) | 0

9. Secondary Outcome: Expression of NKG2 Ligands of Leukemic Blasts
Time Frame: Up to 5 years
Population: Analysis for this endpoint not feasible due to funding constraint.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes